CLINICAL TRIAL: NCT01919164
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Parallel-group Trial to Investigate the Efficacy and Safety of Different Intra Articular (i.a.) Dosages of Sprifermin in Subjects With Primary Osteoarthritis of the Knee
Brief Title: A Study to Investigate the Safety and Effectiveness of Different Doses of Sprifermin in Participants With Osteoarthritis of the Knee
Acronym: FORWARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Nordic Bioscience A/S (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR700692_006; 2011-003059-20 (EudraCT Number)
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis of knee; Recombinant Human Fibroblast Growth Factor-18 (rhFGF-18); Sprifermin; Placebo
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — fibroblast growth factor 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Participants received Placebo matched to Sprifermin as intra-articular injection once every week for 3 consecutive weeks for 4 cycles, that is at week 0, 1, 2 in Cycle 1; at week 26, 27, 28 in Cycle 2; at week 52, 53, 54 in Cycle 3 and at week 78, 79, 80 in Cycle 4 at interval of 6 months.
  Interventions: Drug: Placebo
- Sprifermin (AS902330) 30 mcg/placebo - 2 Cycles (Experimental): Participants received Sprifermin 30 mcg as intra-articular injection once every week for 3 consecutive weeks for 2 alternative cycles, that is at week 0, 1, 2 in Cycle 1 and at week 52, 53, 54 in Cycle 3; and received placebo matched to Sprifermin once every week for 3 consecutive weeks for 2 alternative cycles, that is at week 26, 27, 28 in Cycle 2 and at week 78, 79, 80 in Cycle 4 at interval of 6 months.
  Interventions: Drug: Sprifermin; Drug: Placebo
- Sprifermin (AS902330) 30 mcg- 4 Cycles (Experimental): Participants received Sprifermin 30 micrograms (mcg) as intra-articular injection once every week for 3 consecutive weeks for 4 cycles, that is at week 0, 1, 2 in Cycle 1; at week 26, 27, 28 in Cycle 2; at week 52, 53, 54 in Cycle 3 and at week 78, 79, 80 in Cycle 4 at interval of 6 months.
  Interventions: Drug: Sprifermin
- Sprifermin (AS902330) 100 mcg/Placebo (2 cycles) (Experimental): Participants received Sprifermin 100 mcg as intra-articular injection once every week for 3 consecutive weeks for 2 alternative cycles, that is at week 0, 1, 2 in Cycle 1 and at week 52, 53, 54 in Cycle 3; and received placebo matched to Sprifermin once every week for 3 consecutive weeks for 2 alternative cycles, that is at week 26, 27, 28 in Cycle 2 and at week 78, 79, 80 in Cycle 4 at interval of 6 months.
  Interventions: Drug: Sprifermin; Drug: Placebo
- Sprifermin (AS902330) 100 mcg- 4 Cycles (Placebo Comparator): Participants received Sprifermin 100 mcg as intra-articular injection once every week for 3 consecutive weeks for 4 cycles, that is at week 0, 1, 2 in Cycle 1; at week 26, 27, 28 in Cycle 2; at week 52, 53, 54 in Cycle 3 and at week 78, 79, 80 in Cycle 4 at interval of 6 months.
  Interventions: Drug: Sprifermin

INTERVENTIONS:
Drug: Sprifermin — Participants received Sprifermin as intra-articular injection.
  Other Names: Recombinant Human Fibroblast Growth Factor-18 (rhFGF-18)
  Arms: Sprifermin (AS902330) 100 mcg- 4 Cycles; Sprifermin (AS902330) 100 mcg/Placebo (2 cycles); Sprifermin (AS902330) 30 mcg- 4 Cycles; Sprifermin (AS902330) 30 mcg/placebo - 2 Cycles
Drug: Placebo — Participants received Placebo matched to sprifermin as intra-articular injection.
  Arms: Placebo; Sprifermin (AS902330) 100 mcg/Placebo (2 cycles); Sprifermin (AS902330) 30 mcg/placebo - 2 Cycles

SUMMARY:
This was a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase 2 trial of Sprifermin administered intra-articularly in participants with primary osteoarthritis of the knee and Kellgren-Lawrence Grade 2 or 3. The trial was intended to investigate the efficacy and safety of different intra articular dosages of Sprifermin in these individuals.

DETAILED DESCRIPTION:
Participants were equally randomized to either one of 4 treatment arms or a placebo arm. The trial consists of a Screening period lasting up to 42 days, a two-year double-blind placebo-controlled (DBPC) treatment phase, which begins at randomization (Week 0) and ends at Year 2, and a 3-year extended follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 85 years; of either sex
* Primary femorotibial osteoarthritis according to American College of Rheumatology (ACR) clinical and radiographic criteria , and meeting protocol-specified X-ray criteria in the target knee at screening
* Pain score in the target knee and/or the need for regular symptomatic treatment of knee pain with paracetamol (acetaminophen), systemic non-steroidal anti-inflammatory drugs (NSAIDs) including cyclooxygenase (COX)-2 selective inhibitors (coxibs), or tramadol on most days in the previous month (that is, more than half of the days in the previous month)
* A history of pain due to Osteoarthritis in the target knee for at least 6 months
* A protocol-specified pain score for the target knee in response to Question 1 of the WOMAC pain index ("how much pain have you had [in the target knee, over the past 48 hours] when walking on a flat surface?") after washout of at least 5 half-lives of analgesic medication(s): acetaminophen, topical or oral NSAIDS, coxibs, opioids, and/or tramadol
* Women of childbearing potential must use a form of contraception with a failure rate of less than 1 percent per year throughout the trial

Exclusion Criteria:

* Malalignment of greater than 5 degrees in the femorotibial axis of the target knee
* Clinical signs of inflammation (redness) in the target knee
* Intra-articular administration of corticosteroids or hyaluronic acid into either knee within 6 months before Screening
* Planned knee surgery (affecting either the target or the contralateral knee) within the next two years
* Concomitant conditions or treatments deemed to be incompatible with trial participation
* Any contraindication to MRI according to MRI guidelines, including the inability to undergo a knee MRI exam because of inability to fit in the scanner or knee coil
* Pregnancy or breastfeeding
* Participation in another clinical trial within the 30 days (or 5 half-lives of the investigated compound, whichever is longer) before screening
* Legal incapacity or limited legal capacity

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, MD, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (13):
- United States (2):
  - Research site, Lakewood, Colorado
  - Research site, Baltimore, Maryland
- Research site, Buenos Aires, Argentina
- Czechia (3):
  - Research site, Brno
  - Research site, Pardubice
  - Research site, Prague
- Denmark (3):
  - Research site, Aalborg
  - Research site, Ballerup Municipality
  - Research site, Vejle
- Research site, Tallinn, Estonia
- Research Site, Hong Kong, Hong Kong
- Research site, Lodz, Poland
- Research site, Bucharest, Romania

REFERENCES:
- [Derived] Conaghan PG, Katz N, Hunter DJ, Guermazi A, Hochberg MC, Somberg K, Clive J, Knight C, Johnson M, Zhao L, Goel N. Exploring a novel outcome measure of symptom progression in knee osteoarthritis utilizing a large randomized trial. Osteoarthritis Cartilage. 2025 Mar;33(3):383-390. doi: 10.1016/j.joca.2024.12.003. Epub 2024 Dec 28. PMID 39734047
- [Derived] Eckstein F, Maschek S, Wirth W, Ladel C, Bihlet AR, Knight C, Somberg K, Zhao L. Unbiased analysis of knee cartilage thickness change over three years after sprifermin vs. placebo treatment - A post-hoc analysis from the phase 2B FORWARD study. Osteoarthr Cartil Open. 2024 Aug 23;6(4):100513. doi: 10.1016/j.ocarto.2024.100513. eCollection 2024 Dec. PMID 39286575
- [Derived] Eckstein F, Hochberg MC, Guehring H, Moreau F, Ona V, Bihlet AR, Byrjalsen I, Andersen JR, Daelken B, Guenther O, Ladel C, Michaelis M, Conaghan PG. Long-term structural and symptomatic effects of intra-articular sprifermin in patients with knee osteoarthritis: 5-year results from the FORWARD study. Ann Rheum Dis. 2021 Aug;80(8):1062-1069. doi: 10.1136/annrheumdis-2020-219181. Epub 2021 May 7. PMID 33962962
- [Derived] Guehring H, Moreau F, Daelken B, Ladel C, Guenther O, Bihlet AR, Wirth W, Eckstein F, Hochberg M, Conaghan PG. The effects of sprifermin on symptoms and structure in a subgroup at risk of progression in the FORWARD knee osteoarthritis trial. Semin Arthritis Rheum. 2021 Apr;51(2):450-456. doi: 10.1016/j.semarthrit.2021.03.005. Epub 2021 Mar 11. PMID 33752164
- [Derived] Eckstein F, Kraines JL, Aydemir A, Wirth W, Maschek S, Hochberg MC. Intra-articular sprifermin reduces cartilage loss in addition to increasing cartilage gain independent of location in the femorotibial joint: post-hoc analysis of a randomised, placebo-controlled phase II clinical trial. Ann Rheum Dis. 2020 Apr;79(4):525-528. doi: 10.1136/annrheumdis-2019-216453. Epub 2020 Feb 25. PMID 32098758
- [Derived] Hochberg MC, Guermazi A, Guehring H, Aydemir A, Wax S, Fleuranceau-Morel P, Reinstrup Bihlet A, Byrjalsen I, Ragnar Andersen J, Eckstein F. Effect of Intra-Articular Sprifermin vs Placebo on Femorotibial Joint Cartilage Thickness in Patients With Osteoarthritis: The FORWARD Randomized Clinical Trial. JAMA. 2019 Oct 8;322(14):1360-1370. doi: 10.1001/jama.2019.14735. PMID 31593273
- See also: Trial Awareness and Transparency website Scope — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR700692_006
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 549 participants were randomized in this study.
Groups:
- Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles: Participants received Sprifermin 30 micrograms (mcg) as intra-articular injection once every week for 3 consecutive weeks for 2 alternative cycles, that is at week 0, 1, 2 in Cycle 1 and at week 52, 53, 54 in Cycle 3; and received placebo matched to Sprifermin once every week for 3 consecutive weeks for 2 alternative cycles, that is at week 26, 27, 28 in Cycle 2 and at week 78, 79, 80 in Cycle 4 at interval of 6 months.
Period: Overall Study
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Started | 108 | 110 | 111 | 110 | 110
Safety Analysis Set (Arm assignments for participants in Safety Set were based on actual treatment received.) | 107 | 109 (1 participant assigned to Placebo arm who inadvertently received 30 mcg was included in this arm.) | 111 | 111 (1 participant in Sprifermin2 Cycles arm who inadvertently received 100 mcg was included in this arm.) | 109
Completed | 65 | 80 | 74 | 82 | 77
Not Completed | 43 | 30 | 37 | 28 | 33
Not completed — Adverse Event | 6 | 4 | 9 | 3 | 2
Not completed — Lost to Follow-up | 2 | 2 | 2 | 0 | 4
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 6 | 0 | 3 | 2 | 2
Not completed — Disease progression | 2 | 2 | 1 | 2 | 1
Not completed — Withdrew consent | 13 | 13 | 14 | 14 | 9
Not completed — Other Un-specified | 13 | 9 | 8 | 7 | 15

BASELINE CHARACTERISTICS:
Groups:
- Sprifermin (AS902330) 100 mcg/Placebo- 2 Cycles: Participants received Sprifermin 100 mcg as intra-articular injection once every week for 3 consecutive weeks for 2 alternative cycles, that is at week 0, 1, 2 in Cycle 1 and at week 52, 53, 54 in Cycle 3; and received placebo matched to Sprifermin once every week for 3 consecutive weeks for 2 alternative cycles, that is at week 26, 27, 28 in Cycle 2 and at week 78, 79, 80 in Cycle 4 at interval of 6 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo- 2 Cycles | Sprifermin (AS902330) 100 mcg- 4 Cycles | Total
Number analyzed (Participants) | 108 | 110 | 111 | 110 | 110 | 549
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 46 | 52 | 52 | 46 | 250
  >=65 years | 54 | 64 | 59 | 58 | 64 | 299
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 73 | 80 | 77 | 73 | 379
  Male | 32 | 37 | 31 | 33 | 37 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 107 | 109 | 111 | 110 | 110 | 547
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 21 | 22 | 23 | 23 | 21 | 110
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 87 | 88 | 88 | 87 | 89 | 439
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cartilage Thickness in the Total Femorotibial Joint as Evaluated by Quantitative Magnetic Resonance Imaging (qMRI) at Year 2
Description: The change in cartilage thickness at 2 years was calculated based on quantitative magnetic resonance imaging (qMRI).
Time Frame: Baseline, Year 2 (Week 104)
Population: Modified intent to treat (ITT) analysis set included all randomized participants that is, only planned treatment regimen was used and who had a baseline, at least 1 post-treatment qMRI assessment available in double-blind placebo-controlled part. Here "Number of Participants analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 83 | 92 | 83 | 90 | 86
millimeters | -0.02 (0.07) | -0.01 (0.07) | 0.00 (0.07) | 0.02 (0.08) | 0.03 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles; Descriptive statistics was provided for primary endpoint; Test type: Superiority; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.01 to 0.03]
Statistical Analysis 2: Comparison: Placebo vs Sprifermin (AS902330) 30 mcg- 4 Cycles; Descriptive statistics was provided for primary endpoint; Test type: Superiority; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.01 to 0.04]
Statistical Analysis 3: Comparison: Placebo vs Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles); Descriptive statistics was provided for primary endpoint; Test type: Superiority; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [0.02 to 0.06]
Statistical Analysis 4: Comparison: Placebo vs Sprifermin (AS902330) 100 mcg- 4 Cycles; Descriptive statistics was provided for primary endpoint; Test type: Superiority; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0.03 to 0.07]

2. Secondary Outcome: Changes From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale, Stiffness Subscale, Physical Function Subscale and Total Score at Week 52, Week 78 and Week 104
Description: WOMAC pain subscale consists of 5 questions (Likert Scale) relating to pain. Sum of items of pain subscale ranges from 0-11. Higher scores=worse pain. Stiffness subscale consists of 2 questions relating articular function. Sum of items of stiffness subscale ranges from 0-8. Higher scores=worse function. Physical function subscale consists of 17 question relating to physical activities. Sum of items of physical function subscale ranges from 0-68. Higher scores= worse functional limitations. Each sub-scale is directly transformed into a 0-100 scale, where higher score indicates worse condition. WOMAC total score(24questions) is sum of total subscales which was directly transformed into score range from 0-100. Higher scores=worse condition. Negative value in change is indicative of improvement.
Time Frame: Baseline, Week 52, Week 78 and Week 104
Population: Intention-to-Treat (ITT) analysis set included all participants randomly allocated to a treatment, based on the intention to treat "as randomized" principle. Here "Number of Participants analyzed" = participants evaluable for this outcome measure and "Number analyzed" included those who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 94 | 98 | 89 | 98 | 100
score on a scale
  Pain: Change at Week 52: number analyzed (Participants) | 94 | 98 | 87 | 98 | 100
  Pain: Change at Week 52 | -18.51 (19.49) | -21.55 (18.36) | -15.40 (18.31) | -21.12 (19.73) | -23.34 (17.92)
  Pain: Change at Week 78: number analyzed (Participants) | 90 | 94 | 86 | 94 | 94
  Pain: Change at Week 78 | -21.04 (20.81) | -23.00 (20.42) | -18.19 (21.15) | -23.21 (19.42) | -23.23 (18.41)
  Pain: Change at Week 104: number analyzed (Participants) | 86 | 98 | 89 | 96 | 95
  Pain: Change at Week 104 | -25.37 (20.60) | -23.22 (21.42) | -21.42 (21.37) | -23.15 (18.18) | -26.06 (18.39)
  Stiffness: Change at Week 52: number analyzed (Participants) | 94 | 98 | 87 | 98 | 100
  Stiffness: Change at Week 52 | -18.88 (24.72) | -18.52 (22.89) | -11.09 (21.14) | -16.68 (20.93) | -17.35 (22.16)
  Stiffness: Change at Week 78: number analyzed (Participants) | 90 | 98 | 86 | 94 | 94
  Stiffness: Change at Week 78 | -20.44 (26.76) | -19.47 (25.87) | -14.94 (23.66) | -19.63 (20.38) | -21.44 (23.99)
  Stiffness: Change at Week 104: number analyzed (Participants) | 86 | 98 | 89 | 96 | 95
  Stiffness: Change at Week 104 | -23.20 (25.84) | -20.56 (23.93) | -17.75 (22.74) | -17.76 (20.75) | -22.79 (24.60)
  Function: Change at Week 52: number analyzed (Participants) | 94 | 98 | 87 | 98 | 100
  Function: Change at Week 52 | -15.51 (19.14) | -16.84 (17.64) | -12.01 (18.04) | -14.80 (19.07) | -16.91 (19.69)
  Function: Change at Week 78: number analyzed (Participants) | 90 | 94 | 86 | 94 | 94
  Function: Change at Week 78 | -17.38 (21.01) | -18.23 (19.41) | -16.00 (20.82) | -17.51 (18.96) | -19.29 (19.56)
  Function: Change at Week 104 | -20.89 (20.10) | -20.00 (20.99) | -19.06 (21.52) | -17.03 (20.16) | -20.82 (20.39)
  Total: Change at Week 52: number analyzed (Participants) | 94 | 98 | 87 | 98 | 100
  Total: Change at Week 52 | -16.42 (18.61) | -17.97 (16.95) | -12.64 (17.42) | -16.29 (18.35) | -18.29 (18.25)
  Total: Change at Week 78: number analyzed (Participants) | 90 | 94 | 86 | 94 | 94
  Total: Change at Week 78 | -18.41 (20.43) | -19.34 (19.15) | -16.36 (20.35) | -18.88 (18.15) | -20.29 (18.49)
  Total: Change at Week 104: number analyzed (Participants) | 86 | 98 | 89 | 96 | 95
  Total: Change at Week 104 | -22.02 (19.70) | -20.73 (20.22) | -19.44 (20.88) | -18.37 (18.69) | -22.08 (19.11)

3. Secondary Outcome: Change From Baseline in the 20-meter Walk Test at Week 12, 26, 38, 52, 64, 78, 90 and 104
Description: The 20-meter walk test is an objective test of physical function which consists of measuring the time needed for the participant to walk 20 meters at a normal pace. A stopwatch was used for time measurement.
Time Frame: Baseline, Week 12, 26, 38, 52, 64, 78, 90 and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 105 | 108 | 109 | 107 | 108
seconds
  Change at Week 12 | -1.2 (2.9) | -0.4 (4.0) | -0.5 (2.6) | -0.8 (2.2) | -1.1 (3.3)
  Change at Week 26: number analyzed (Participants) | 99 | 108 | 101 | 103 | 102
  Change at Week 26 | -1.3 (3.7) | -0.4 (3.9) | -0.3 (2.6) | -1.1 (2.8) | -1.3 (3.0)
  Change at Week 38: number analyzed (Participants) | 98 | 103 | 98 | 102 | 98
  Change at Week 38 | -1.1 (3.6) | -0.5 (3.4) | -0.7 (2.5) | -1.0 (2.9) | -1.4 (3.2)
  Change at Week 52: number analyzed (Participants) | 95 | 101 | 90 | 101 | 100
  Change at Week 52 | -1.7 (4.2) | -1.1 (3.6) | -0.7 (2.5) | -0.4 (7.9) | -1.3 (2.8)
  Change at Week 64: number analyzed (Participants) | 92 | 101 | 93 | 97 | 93
  Change at Week 64 | -1.8 (3.6) | -1.5 (4.1) | -0.9 (2.5) | -1.3 (2.6) | -1.6 (3.4)
  Change at Week 78: number analyzed (Participants) | 91 | 96 | 88 | 97 | 94
  Change at Week 78 | -1.6 (3.7) | -1.0 (4.0) | -0.8 (2.8) | -1.6 (3.0) | -1.3 (3.2)
  Change at Week 90: number analyzed (Participants) | 83 | 96 | 87 | 91 | 87
  Change at Week 90 | -2.1 (3.9) | -1.0 (3.2) | -1.1 (2.7) | -1.8 (3.1) | -1.7 (3.5)
  Change at Week 104: number analyzed (Participants) | 87 | 100 | 91 | 99 | 94
  Change at Week 104 | -1.6 (4.0) | -1.2 (4.1) | -0.8 (3.4) | -1.4 (2.9) | -1.3 (3.2)

4. Secondary Outcome: Change From Baseline in the Patient's Global Assessment (PGA) at Week 12, 26, 38, 52, 64, 78, 90 and 104
Description: The Patient Global Assessment is based on participant's answer to the question "Considering all the ways your osteoarthritis of the knee has affected you during the last 48 Hours, select the number that best describes the impact of your knee osteoarthritis on your daily life", and can take on values between 0-10 (0=None, 10=Extreme), for summaries the values are rescaled to 0-100 by multiplication with 10. Higher scores indicated worsening of condition. A negative value in change in Patient's Global Assessment is indicative of an improvement.
Time Frame: Baseline, Week 12, 26, 38, 52, 64, 78, 90 and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 104 | 108 | 109 | 106 | 107
score on a scale
  Change at Week 12 | -16.6 (23.5) | -13.9 (20.6) | -17.0 (25.0) | -15.0 (23.2) | -16.7 (22.1)
  Change at Week 26: number analyzed (Participants) | 99 | 108 | 100 | 103 | 102
  Change at Week 26 | -16.3 (22.3) | -15.1 (22.7) | -17.7 (25.3) | -18.7 (22.4) | -19.1 (24.1)
  Change at Week 38: number analyzed (Participants) | 98 | 103 | 97 | 102 | 98
  Change at Week 38 | -18.9 (26.2) | -17.2 (22.5) | -19.2 (24.9) | -20.5 (24.3) | -18.4 (25.1)
  Change at Week 52: number analyzed (Participants) | 95 | 100 | 88 | 101 | 100
  Change at Week 52 | -19.6 (25.8) | -20.9 (21.2) | -18.0 (23.9) | -19.5 (25.2) | -21.6 (24.0)
  Change at Week 64: number analyzed (Participants) | 92 | 101 | 93 | 97 | 93
  Change at Week 64 | -22.7 (24.6) | -21.7 (21.9) | -22.3 (23.0) | -21.6 (25.8) | -21.3 (24.6)
  Change at Week 78: number analyzed (Participants) | 91 | 96 | 88 | 97 | 93
  Change at Week 78 | -22.7 (26.5) | -21.5 (24.1) | -23.1 (25.7) | -22.0 (25.4) | -24.2 (24.1)
  Change at Week 90: number analyzed (Participants) | 83 | 97 | 87 | 91 | 87
  Change at Week 90 | -25.8 (25.6) | -22.3 (24.5) | -21.7 (24.8) | -21.1 (26.3) | -26.2 (24.9)
  Change at Week 104: number analyzed (Participants) | 87 | 100 | 91 | 99 | 95
  Change at Week 104 | -27.5 (25.0) | -23.0 (22.3) | -23.8 (24.9) | -22.1 (25.6) | -25.8 (22.8)

5. Secondary Outcome: Change From Baseline in Minimal Joint Space Width (mJSW) in the Medial and Lateral Compartments as Evaluated by X-ray at Week 52 and 104
Description: Change in joint space narrowing was visualized with the "fixed flexion" knee radiograph. Determination of joint space narrowing by X-ray is considered to be a semi-quantitative method for assessment of progression of knee Osteoarthritis (OA). X-rays of both the target knee and the contralateral knee were performed. X-rays were read centrally. X-ray images were used to measure mJSW in the medial femorotibial and lateral femorotibial compartments and to determine the participant's baseline Kellgren-Lawrence grades (KLG).
Time Frame: Baseline, Week 52 and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 95 | 101 | 95 | 100 | 101
millimeter
  Medial: Change at Week 52: number analyzed (Participants) | 95 | 97 | 89 | 100 | 101
  Medial: Change at Week 52 | -0.10 (0.48) | -0.05 (0.53) | -0.04 (0.43) | 0.02 (0.55) | -0.04 (0.57)
  Medial: Change at Week 104: number analyzed (Participants) | 90 | 101 | 95 | 98 | 95
  Medial: Change at Week 104 | -0.11 (0.59) | -0.09 (0.73) | 0.03 (0.52) | -0.05 (0.66) | -0.07 (0.86)
  Lateral: Change at Week 52: number analyzed (Participants) | 95 | 97 | 89 | 100 | 101
  Lateral: Change at Week 52 | 0.07 (0.46) | -0.03 (0.62) | 0.16 (0.54) | 0.10 (0.37) | 0.14 (0.43)
  Lateral: Change at Week 104: number analyzed (Participants) | 90 | 101 | 95 | 98 | 95
  Lateral: Change at Week 104 | -0.07 (0.49) | -0.03 (0.64) | 0.01 (0.65) | 0.19 (0.49) | 0.19 (0.49)

6. Secondary Outcome: Change From Baseline in Cartilage Thickness in the Medial and Lateral Compartments as Well as in the Total Femorotibial Joint
Description: The change in cartilage thickness was calculated based on quantitative magnetic resonance imaging (qMRI).
Time Frame: Medial and Lateral: Baseline, Week 26, 52, 78 and 104; Total: Baseline, Week 26, 52 and 78
Population: Modified ITT analysis set was used. Here "Number of Participants analyzed" = participants evaluable for this outcome measure and "Number analyzed" included those who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 94 | 97 | 97 | 96 | 99
millimeter
  Medial: Change at Week 26: number analyzed (Participants) | 93 | 97 | 95 | 95 | 99
  Medial: Change at Week 26 | 0.00 (0.06) | 0.00 (0.06) | -0.01 (0.06) | 0.01 (0.05) | 0.01 (0.06)
  Medial: Change at Week 52: number analyzed (Participants) | 91 | 93 | 81 | 94 | 93
  Medial: Change at Week 52 | -0.01 (0.06) | -0.01 (0.07) | -0.01 (0.06) | 0.00 (0.07) | 0.01 (0.06)
  Medial: Change at Week 78: number analyzed (Participants) | 84 | 91 | 84 | 90 | 89
  Medial: Change at Week 78 | -0.01 (0.07) | -0.01 (0.07) | 0.01 (0.06) | 0.01 (0.10) | 0.03 (0.08)
  Medial: Change at Week 104: number analyzed (Participants) | 83 | 92 | 83 | 90 | 86
  Medial: Change at Week 104 | -0.03 (0.12) | -0.02 (0.10) | -0.01 (0.08) | 0.00 (0.11) | 0.02 (0.08)
  Lateral: Change at Week 26 | -0.01 (0.05) | 0.00 (0.05) | 0.00 (0.06) | 0.02 (0.05) | 0.02 (0.05)
  Lateral: Change at Week 52: number analyzed (Participants) | 92 | 93 | 83 | 95 | 93
  Lateral: Change at Week 52 | -0.01 (0.05) | -0.01 (0.07) | 0.00 (0.05) | 0.02 (0.06) | 0.02 (0.05)
  Lateral: Change at Week 78: number analyzed (Participants) | 85 | 91 | 85 | 91 | 89
  Lateral: Change at Week 78 | 0.00 (0.05) | 0.01 (0.06) | 0.01 (0.08) | 0.03 (0.07) | 0.03 (0.06)
  Lateral: Change at Week 104: number analyzed (Participants) | 83 | 92 | 85 | 91 | 86
  Lateral: Change at Week 104 | -0.01 (0.05) | -0.01 (0.07) | 0.00 (0.09) | 0.04 (0.07) | 0.04 (0.06)
  Total: Change at Week 26: number analyzed (Participants) | 93 | 97 | 95 | 95 | 99
  Total: Change at Week 26 | -0.01 (0.05) | 0.00 (0.04) | 0.00 (0.05) | 0.01 (0.04) | 0.01 (0.05)
  Total: Change at Week 52: number analyzed (Participants) | 91 | 93 | 81 | 94 | 93
  Total: Change at Week 52 | -0.01 (0.05) | -0.01 (0.06) | 0.00 (0.05) | 0.01 (0.06) | 0.01 (0.05)
  Total: Change at Week 78: number analyzed (Participants) | 84 | 91 | 84 | 90 | 89
  Total: Change at Week 78 | -0.01 (0.05) | 0.00 (0.06) | 0.06 (0.06) | 0.02 (0.07) | 0.03 (0.06)

7. Secondary Outcome: Change From Baseline in Cartilage-Volume in the Medial and Lateral Compartments as Well as in the Total Femorotibial Joint at Week 26, 52, 78 and 104
Description: The change in cartilage volume in the medial and lateral compartments as well as in the total femorotibial joint at Week 26, 52, 78 and 104 was calculated based on qMRI.
Time Frame: Baseline, Week 26, 52, 78 and 104
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: microliter
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 94 | 97 | 97 | 96 | 99
microliter
  Medial: Change at Week 26: number analyzed (Participants) | 93 | 97 | 95 | 95 | 99
  Medial: Change at Week 26 | 0.0 (112.2) | 1.7 (110.8) | -3.2 (99.5) | 16.7 (89.8) | 16.5 (114.2)
  Medial: Change at Week 52: number analyzed (Participants) | 91 | 93 | 81 | 94 | 93
  Medial: Change at Week 52 | -10.2 (100.7) | -2.9 (127.1) | -7.0 (103.7) | 3.6 (127.5) | 16.5 (110.6)
  Medial: Change at Week 78: number analyzed (Participants) | 84 | 91 | 84 | 90 | 89
  Medial: Change at Week 78 | -8.9 (125.3) | -7.0 (153.7) | 23.6 (109.3) | 33.2 (177.0) | 53.9 (147.3)
  Medial: Change at Week 104: number analyzed (Participants) | 83 | 92 | 83 | 90 | 86
  Medial: Change at Week 104 | -41.0 (192.1) | -21.4 (198.3) | 3.6 (123.9) | 19.5 (202.3) | 48.6 (150.7)
  Lateral: Change at Week 26 | -12.8 (84.4) | 0.8 (82.0) | 1.5 (102.3) | 31.3 (87.7) | 25.1 (85.8)
  Lateral: Change at Week 52: number analyzed (Participants) | 92 | 93 | 83 | 95 | 93
  Lateral: Change at Week 52 | -12.7 (94.0) | -17.5 (141.1) | 2.7 (98.2) | 32.4 (107.5) | 28.1 (87.3)
  Lateral: Change at Week 78: number analyzed (Participants) | 85 | 91 | 85 | 91 | 89
  Lateral: Change at Week 78 | -1.8 (89.7) | 13.9 (113.6) | 21.6 (129.0) | 55.9 (123.1) | 55.2 (101.6)
  Lateral: Change at Week 104: number analyzed (Participants) | 83 | 92 | 85 | 91 | 86
  Lateral: Change at Week 104 | -14.5 (87.2) | -6.8 (144.9) | 7.2 (134.8) | 75.5 (111.8) | 67.9 (112.5)
  Total: Change at Week 26: number analyzed (Participants) | 93 | 97 | 95 | 95 | 99
  Total: Change at Week 26 | -13.0 (163.2) | 2.5 (147.0) | -2.9 (161.8) | 48.4 (150.9) | 41.5 (166.6)
  Total: Change at Week 52: number analyzed (Participants) | 91 | 93 | 81 | 94 | 93
  Total: Change at Week 52 | -23.7 (155.7) | -20.4 (217.6) | -5.5 (169.0) | 36.2 (203.1) | 44.7 (163.2)
  Total: Change at Week 78: number analyzed (Participants) | 84 | 91 | 84 | 90 | 89
  Total: Change at Week 78 | -10.3 (176.8) | 6.9 (228.1) | 44.8 (195.3) | 89.9 (272.6) | 109.1 (219.1)
  Total: Change at Week 104: number analyzed (Participants) | 83 | 92 | 83 | 90 | 86
  Total: Change at Week 104 | -55.5 (239.5) | -28.2 (275.7) | 9.5 (205.7) | 96.6 (271.1) | 116.5 (233.5)

8. Secondary Outcome: Synovial Fluid Levels of Sprifermin/FGF-18
Description: Levels of sprifermin/FGF-18 in synovial fluid were measured to provide a first estimate of the residence time of sprifermin in the synovial fluid.
Time Frame: Pre-dose at Week 0, 2 hours post-dose at Week 1 and 2 of Cycle 1, 2, 3 and 4 (each cycle is of 28 days)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Arm assignments for participants in Safety Set were based on actual treatment received. Here "Number of Participants analyzed" = participants evaluable for this outcome measure and "Number analyzed" are those who were evaluable at specified timepoint.
Measure: Median (Full Range); unit: picogram/milliliter
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 3 | 20 | 22 | 25 | 27
picogram/milliliter
  Week 0; Cycle 1: number analyzed (Participants) | 0 | 5 | 5 | 5 | 8
  Week 0; Cycle 1 |  | 56876.4 [5843.8 to 86068.0] | 1006.5 [206.6 to 34439.4] | 1386.1 [260.4 to 36766.4] | 5896.4 [631.3 to 238780.1]
  Week 1; Cycle 1: number analyzed (Participants) | 2 | 5 | 7 | 10 | 16
  Week 1; Cycle 1 | 622.1 [156.0 to 1088.2] | 3628.3 [229.9 to 37140.5] | 1493.2 [214.2 to 110515.4] | 359.8 [151.2 to 37014.8] | 1062.3 [156.7 to 840122.2]
  Week 2; Cycle 1: number analyzed (Participants) | 0 | 10 | 6 | 12 | 16
  Week 2; Cycle 1 |  | 3150.9 [189.1 to 33378.5] | 4167.0 [460.3 to 8857.1] | 467.9 [150.7 to 108866.0] | 258.2 [171.9 to 48066.3]
  Week 0; Cycle 2: number analyzed (Participants) | 1 | 0 | 10 | 1 | 13
  Week 0; Cycle 2 | 202.5 [202.5 to 202.5] |  | 7039.1 [309.8 to 1108182.4] | 308.2 [308.2 to 308.2] | 32360.2 [559.9 to 683691.9]
  Week 1; Cycle 2: number analyzed (Participants) | 0 | 0 | 17 | 0 | 16
  Week 1; Cycle 2 |  |  | 14756.3 [904.6 to 359059.2] |  | 7036.9 [159.9 to 82301.6]
  Week 2; Cycle 2: number analyzed (Participants) | 0 | 0 | 16 | 0 | 18
  Week 2; Cycle 2 |  |  | 6408.3 [154.4 to 220629.5] |  | 1146.7 [156.1 to 42598.5]
  Week 0; Cycle 3: number analyzed (Participants) | 3 | 20 | 15 | 9 | 13
  Week 0; Cycle 3 | 463.7 [223.8 to 5386.5] | 8019.3 [279.2 to 358231.4] | 9443.4 [505.7 to 271320.6] | 16901.2 [461.0 to 273247.0] | 20753.0 [4119.1 to 303440.5]
  Week 1; Cycle 3: number analyzed (Participants) | 0 | 14 | 11 | 16 | 22
  Week 1; Cycle 3 |  | 8607.6 [276.7 to 147723.9] | 4605.1 [337.2 to 358029.6] | 3908.8 [177.5 to 86823.9] | 10160.0 [165.5 to 375638.7]
  Week 2; Cycle 3: number analyzed (Participants) | 1 | 15 | 15 | 25 | 25
  Week 2; Cycle 3 | 260.9 [260.9 to 260.9] | 9592.2 [1277.1 to 35615.5] | 9422.2 [409.3 to 353582.4] | 1801.0 [171.9 to 77338.9] | 4161.7 [151.1 to 213692.3]
  Week 0; Cycle 4: number analyzed (Participants) | 0 | 0 | 17 | 0 | 16
  Week 0; Cycle 4 |  |  | 12458.4 [224.6 to 163129.3] |  | 22132.1 [215.7 to 897758.2]
  Week 1; Cycle 4: number analyzed (Participants) | 1 | 0 | 18 | 1 | 22
  Week 1; Cycle 4 | 215.3 [215.3 to 215.3] |  | 9602.7 [178.6 to 45631.9] | 2285.2 [2285.2 to 2285.2] | 11468.3 [157.5 to 142318.7]
  Week 2; Cycle 4: number analyzed (Participants) | 1 | 0 | 22 | 2 | 27
  Week 2; Cycle 4 | 10670.0 [10670.0 to 10670.0] |  | 7103.8 [196.8 to 384511.5] | 331.1 [168.4 to 493.7] | 8026.4 [179.7 to 272804.6]

9. Secondary Outcome: Serum Levels of Sprifermin/FGF-18
Time Frame: Pre-dose at Week 0, 2 hours post-dose at Week 1 and 2 of Cycle 1, 2, 3 and 4 (each cycle is of 28 days)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Arm assignments for participants in Safety Set were based on actual treatment received.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
Number analyzed (Participants) | 107 | 109 | 111 | 111 | 109
picogram/milliliter | NA (NA) — Serum levels of AS902330/FGF-18 could not be analyzed because the serum concentrations were not quantifiable, as serum sprifermin concentrations were below Lower Limit of Quantification (LLOQ). LLOQ=100 picogram/milliliter. | NA (NA) — Serum levels of AS902330/FGF-18 could not be analyzed because the serum concentrations were not quantifiable, as serum sprifermin concentrations were below Lower Limit of Quantification (LLOQ). LLOQ=100 picogram/milliliter. | NA (NA) — Serum levels of AS902330/FGF-18 could not be analyzed because the serum concentrations were not quantifiable, as serum sprifermin concentrations were below Lower Limit of Quantification (LLOQ). LLOQ=100 picogram/milliliter. | NA (NA) — Serum levels of AS902330/FGF-18 could not be analyzed because the serum concentrations were not quantifiable, as serum sprifermin concentrations were below Lower Limit of Quantification (LLOQ). LLOQ=100 picogram/milliliter. | NA (NA) — Serum levels of AS902330/FGF-18 could not be analyzed because the serum concentrations were not quantifiable, as serum sprifermin concentrations were below Lower Limit of Quantification (LLOQ). LLOQ=100 picogram/milliliter.

ADVERSE EVENTS:
Time Frame: Baseline up to 5 years. Participants were assessed for adverse events for the entire study.
Description: Adverse events are presented as per Safety Set.Arm assignments for participants in Safety Set were based on actual treatment received, such that 1participant assigned to Placebo arm who inadvertently received 30 mcg was included in Sprifermin 30mcg/placebo-2 Cycles arm for purpose of safety analysis. Similarly, 1 participant assigned to Sprifermin 30mcg/placebo-2 Cycles arm who inadvertently received 100 mcg was included in Sprifermin 100mcg/placebo-2 Cycles arm for purpose of safety analysis.
Arm/Group | Placebo | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles | Sprifermin (AS902330) 30 mcg- 4 Cycles | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) | Sprifermin (AS902330) 100 mcg- 4 Cycles
All-Cause Mortality (participants affected / at risk) | 1/107 | 0/109 | 0/111 | 0/111 | 0/109
Serious Adverse Events (participants affected / at risk) | 39/107 | 35/109 | 34/111 | 32/111 | 41/109
Other Adverse Events (participants affected / at risk) | 105/107 | 106/109 | 109/111 | 106/111 | 107/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=107) | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles (N=109) | Sprifermin (AS902330) 30 mcg- 4 Cycles (N=111) | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) (N=111) | Sprifermin (AS902330) 100 mcg- 4 Cycles (N=109)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 1 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 4 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 10 | 7 | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Arachnoid cyst (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrom (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Meningeal disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Removal of internal fixation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 2
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=107) | Sprifermin (AS902330) 30 mcg/Placebo - 2 Cycles (N=109) | Sprifermin (AS902330) 30 mcg- 4 Cycles (N=111) | Sprifermin (AS902330) 100 mcg/Placebo (2 Cycles) (N=111) | Sprifermin (AS902330) 100 mcg- 4 Cycles (N=109)
Hypothyroidism (Endocrine disorders) | 2 | 1 | 1 | 6 | 2
Cataract (Eye disorders) | 8 | 6 | 10 | 6 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 3 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 4 | 8 | 5
Gastritis (Gastrointestinal disorders) | 4 | 4 | 4 | 4 | 6
Toothache (Gastrointestinal disorders) | 5 | 2 | 4 | 7 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 7 | 2 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 2 | 6 | 2
Injection site pain (General disorders) | 6 | 5 | 10 | 4 | 8
Injection site bruising (General disorders) | 4 | 5 | 6 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 21 | 25 | 28 | 28 | 30
Nasopharyngitis (Infections and infestations) | 27 | 25 | 20 | 19 | 22
Urinary tract infection (Infections and infestations) | 10 | 13 | 10 | 13 | 17
Influenza (Infections and infestations) | 13 | 10 | 11 | 12 | 12
Cystitis (Infections and infestations) | 7 | 15 | 8 | 9 | 10
Bronchitis (Infections and infestations) | 10 | 11 | 6 | 6 | 9
Pneumonia (Infections and infestations) | 6 | 9 | 7 | 6 | 3
Viral infection (Infections and infestations) | 5 | 6 | 4 | 4 | 4
Gastroenteritis (Infections and infestations) | 0 | 3 | 7 | 7 | 2
Herpes zoster (Infections and infestations) | 3 | 5 | 2 | 3 | 6
Procedural pain (Injury, poisoning and procedural complications) | 18 | 9 | 9 | 9 | 7
Contusion (Injury, poisoning and procedural complications) | 5 | 9 | 9 | 4 | 9
Ligament sprain (Injury, poisoning and procedural complications) | 6 | 5 | 6 | 2 | 8
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 5 | 7 | 6 | 7
C-reactive protein increased (Investigations) | 3 | 2 | 0 | 3 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 5 | 3 | 10 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 7 | 4 | 6 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 6 | 3 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 58 | 59 | 57 | 55 | 54
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 28 | 29 | 33 | 27
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 | 22 | 24 | 17 | 17
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 16 | 18 | 21 | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 12 | 24 | 18 | 20
Joint swelling (Musculoskeletal and connective tissue disorders) | 10 | 14 | 11 | 12 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 9 | 9 | 7
Spinal pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 5 | 6 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 4 | 4 | 1 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8 | 3 | 6
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 | 8 | 5 | 5 | 4
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 3 | 6 | 7 | 4 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 8 | 2 | 4 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 6 | 3
Headache (Nervous system disorders) | 15 | 14 | 11 | 13 | 18
Sciatica (Nervous system disorders) | 11 | 8 | 4 | 7 | 7
Dizziness (Nervous system disorders) | 7 | 3 | 3 | 5 | 10
Hypoaesthesia (Nervous system disorders) | 7 | 4 | 5 | 3 | 3
Memory impairment (Nervous system disorders) | 4 | 0 | 6 | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 0 | 7 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 12 | 12 | 6 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1 | 2 | 3
Hypertension (Vascular disorders) | 17 | 24 | 14 | 20 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-03-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT01919164/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT01919164/SAP_001.pdf